CLINICAL TRIAL: NCT01632384
Title: The Effects of Smoking Withdrawal on Resting State Functional Connectivity
Acronym: SmokeAtt04
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study close-out
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00031550; R01DA023516 (NIH)
Record Dates: First submitted 2012-02-20; First posted 2012-07-02 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Smoking
Keywords: Smoker; Non-Smoker; Healthy; Drug free; MRI
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Abstain from smoking for 24 hours — Compare smoking satiation to 24 hour smoking abstinence

SUMMARY:
The purpose of this study is to see how the brain differs between smoking regularly and after not smoking for 24 hours. The investigators will be using an MRI machine to get the information from adult smokers and non-smokers while they lie in the scanner with their eyes closed. Smokers will be scanned when they have not smoked for 24 hrs and shortly after smoking. It is our hypothesis that brain activity will be altered after not smoking for 24 hours.

DETAILED DESCRIPTION:
The broad objective of this proposal is to identify functional neuroanatomical correlates of changes in brain functional connectivity during smoking abstinence. The investigators will measure changes in regional blood oxygenation levels using fMRI while adult smokers and non-smokers lie in the scanner with their eyes closed. Smokers will be scanned when they are abstinent from smoking for 24 hrs and shortly after smoking. Our primary hypothesis is that smoking abstinence will alter resting state brain activity (or resting state functional connectivity; RSFC) across widely distributed neural networks and that high-resolution fMRI will help in resolving the exact nature of such changes. Data will be analyzed using methods developed in our laboratory and applied to other resting state datasets. All of the procedures used in the study are well validated and introduce only minor risk to participants (e.g. blood draw; MRI).

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* Drug free
* No known health problems
* Currently not taking any medication
* Uninterested in quitting smoking long term

Exclusion Criteria:

* Left handed/ambidextrous
* Currently taking medication
* Interested in quitting long term

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Blood-oxygen-level-dependent (BOLD) signal | following smoking cigarette 30 minutes prior to scan
  Smokers will be scanned after smoking to satiety. In order to be considered satiated, smokers will have to be regular smokers (smoking daily for at least 2 years).

SECONDARY OUTCOMES:
Blood-oxygen-level-dependent (BOLD) signal | 24 hours abstinence
  Smokers will be asked to stop smoking 24 hours prior to the scan without the aid of nicotine replacement therapies. They will resume smoking as usual 24 hours after the scan.

CONTACTS AND LOCATIONS:
Overall Officials: Francis J McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Health Behavior Neuroscience Research Program, Durham, North Carolina, United States